CLINICAL TRIAL: NCT00491569
Title: NMDA Enhancers in the Treatment of Schizophrenia: Sarcosine vs. D-Serine
Brief Title: Sarcosine or D-Serine Add-on Treatment for Chronic Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); National Health Research Institutes, Taiwan (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NSC-94-2314-B-039-026
Record Dates: First submitted 2007-06-24; First posted 2007-06-26 (Estimated); Last update posted 2007-06-26 (Estimated); Status verified 2007-06

CONDITIONS: Schizophrenias; Psychoses; Psychotic Disorders; Schizophrenic Disorders
Keywords: Schizophrenia; sarcosine; D-serine; NMDA
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Sarcosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sarcosine and D-serine

SUMMARY:
Both GlyT-1 inhibitors and NMDA-glycine site agonists have been demonstrated to be beneficial for chronic schizophrenia patients.

The purpose of this study is to compare efficacy and safety of add-on treatment of sarcosine, a GlyT-1 inhibitor, and D-serine, an NMDA-glycine site agonist, in chronically stable schizophrenia patients who have been stabilized with antipsychotics.

DETAILED DESCRIPTION:
The etiology of schizophrenia remains unclear. Schizophrenia patients reveal positive symptoms, negative symptoms, and cognitive impairments. In addition to dopamine system hyperactivity, hypofunction of N-methyl-D-aspartate (NMDA) receptor plays a role in the pathophysiology of schizophrenia. Consequently, enhancing NMDA receptor neurotransmission has been regarded as a novel treatment approach. To date, there have been several reported trials on NMDA enhancers. Both sarcosine (N-methylglycine, a glycine transporter I inhibitor) and D-serine (a potent NMDA-glycine site agonist) showed therapeutic effects in chronically stable patients. Interestingly, sarcosine appeared more efficacious than D-serine in acutely exacerbated ones when added-on to antipsychotics. Both sarcosine and D-serine yielded excellent safety profiles.

It remains unclear whether sarcosine can be also more efficacious than D-serine in the treatment for chronically stable schizophrenia. The aim of this project is to examine the efficacy and safety of add-on treatment of sarcosine vs. D-serine in chronically stable schizophrenia patients who have been stabilized with antipsychotics.

In the study, 60-75 schizophrenic patients are recruited into the 6-week trial and randomly assigned into the three groups (2 gm/d sarcosine, 2 gm/d D-serine, or placebo) with a double-blind manner. Clinical manifestation (Positive and Negative Syndrome Scale [PANSS], side effects and quality of life (QOL) are evaluated every two weeks during the trial.. The efficacies of three groups are compared.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill the criteria of schizophrenia according to the Diagnostic and Statistic Manual, fourth edition (DSM-IV).
* Agree to participate in the study and provide informed consent.

Exclusion Criteria:

* Meet DSM-IV criteria of major mood disorder, current substance dependence or mental retardation
* History of epilepsy, head trauma or CNS diseases
* Major, untreated medical diseases
* Pregnancy or lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-01; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Total scores of Positive and Negative Syndrome Scale (PANSS) and Quality of Life (QOL) | 6 weeks

SECONDARY OUTCOMES:
Subscales of PANSS | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Yuan Lane, MD,PhD, Principal Investigator — Department of Psychiatry, China Medical University Hospital, Taiwan
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

REFERENCES:
- [Background] Lane HY, Chang YC, Liu YC, Chiu CC, Tsai GE. Sarcosine or D-serine add-on treatment for acute exacerbation of schizophrenia: a randomized, double-blind, placebo-controlled study. Arch Gen Psychiatry. 2005 Nov;62(11):1196-204. doi: 10.1001/archpsyc.62.11.1196. PMID 16275807
- [Derived] Lane HY, Lin CH, Huang YJ, Liao CH, Chang YC, Tsai GE. A randomized, double-blind, placebo-controlled comparison study of sarcosine (N-methylglycine) and D-serine add-on treatment for schizophrenia. Int J Neuropsychopharmacol. 2010 May;13(4):451-60. doi: 10.1017/S1461145709990939. Epub 2009 Nov 4. PMID 19887019